CLINICAL TRIAL: NCT03234439
Title: Digital Tools for Coping With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MyStrength, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017/06/13
Record Dates: First submitted 2017-07-24; First posted 2017-07-31 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pain; Depression; Anxiety; Opioid Use
Keywords: digital behavioral health
MeSH Terms: conditions — Chronic Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Double-arm, waitlist control trail with 1:1 randomization
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myStrength Intervention (Experimental): The myStrength intervention arm will be encouraged to utilize the chronic pain offering consisting of 6 modules. Each module has 5 activities and can take on average 5-15 minutes to complete. Study participants assigned to the myStrength intervention will have one week to complete each module. In addition to completing the required chronic pain modules, study participants in the myStrength intervention arm will have the option to also select other areas of interest and complete corresponding activities at their own pace. myStrength utilization will be recorded and analyzed.
  Interventions: Behavioral: myStrength
- Waitlist Control (No Intervention): The waitlist control group will gain access to the myStrength platform 60 days following the start of the study.

INTERVENTIONS:
Behavioral: myStrength — myStrength is a digital self-care behavioral and wellness platform
  Arms: myStrength Intervention

SUMMARY:
Chronic pain is becoming increasingly more prevalent worldwide. High rates of co-morbid psychological distress are also commonly found among individuals living with chronic pain. Often requiring a multi-modal treatment approach, a growing body of literature suggests that digital behavioral health interventions and tools may serve as promising complementary options to help individuals cope with the pain.

DETAILED DESCRIPTION:
The research objective is to evaluate the effectiveness of the myStrength product offerings, namely the chronic pain focus area, on study participants' functional well-being over time. The research questions to be answered include the following:

1. Do study participants who are randomized to the myStrength intervention arm experience change in their self-reported ability to function, outlook on pain, and/or perception of prescription opioids.
2. Do study participants who are randomized to the myStrength intervention arm experience change in terms of their behavioral health, such as anxiety and depression levels, during the study period.

The study team hypothesizes that myStrength study participants will achieve a higher level of functioning and adopt a more positive outlook toward their pain management as compared to the waitlist control group. Self-assessments will be repeated throughout the study period to capture the inflection point of change as well as the sustainability of these changes over time.

ELIGIBILITY:
Inclusion Criteria:

1. Study participants must be 18 years of age or older
2. Self-report chronic pain lasting for at least the past 3 months but no more than 9 months (examples include lower back pain, arthritis, chronic headaches, neuropathic pain, knee pain)
3. Must have considered, have a history of, or are currently taking a prescription opioid for chronic pain (examples oxycodone (OxyContin, Percodan, Percocet), hydrocodone (Vicodin, Lortab, Lorcet), morphine (Kadian, Avinza, MS Contin), fentanyl (Duragesic), propoxyphene (Darvon), hydromorphone (Dilaudid)
4. Fluent in English and articulate Access to a laptop or mobile device to access email and the myStrength platform

Exclusion Criteria:

1. Under the age of 18
2. Chronic pain due to cancer
3. Chronic pain <3 months or > 9 months
4. Prior exposure to the myStrength platform
5. Self-reported history of hospitalization for mental illness or a substance use disorder
6. Receiving government benefits related to a developmental or behavioral health disability

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in baseline thoughts and feelings about chronic pain as measured by Global Pain Scale at 6 months | Repeated measures over time: baseline and day 180
  Measure ability to function in the presence of chronic pain

SECONDARY OUTCOMES:
Change in baseline PHQ9 at 6 months | Repeated measures over time: baseline and day 180
  Measure self-reported depression symptoms
Change in baseline Current Opioid Misuse Measure at 6 months | Repeated measures over time: baseline and day 180
  Screen for maladaptive opioid use
Change in baseline confidence to live with chronic pain as measured by Pain Self-Efficacy Scale at 6 months | Repeated measures over time: baseline and day 180
  Measure ability to function in the presence of chronic pain
Change in baseline and GAD7 at 6 months | Repeated measures over time: baseline and day 180
  Measure self-reported anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Krista Schladweiler, PhD, Principal Investigator — MyStrength, Inc.
Locations (12):
- United States (12):
  - Craigslist, Los Angeles, California
  - Craigslist, San Francisco, California
  - Craigslist, Denver, Colorado
  - Craigslist, Washington D.C., District of Columbia
  - Craigslist, Miami, Florida
  - Craigslist, Atlanta, Georgia
  - Craigslist, Boston, Massachusetts
  - Craigslist, Minneapolis, Minnesota
  - Craigslist, New York, New York
  - Craigslist, Philadelphia, Pennsylvania
  - Craigslist, Houston, Texas
  - Craigslist, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No